CLINICAL TRIAL: NCT06841900
Title: Implementation of the International Classification of Functioning, Disability and Health Model in Paediatric Cochlear Implant Recipients: a Multi-center Prospective Follow-up Cohort Study
Brief Title: Implementation of the International Classification of Functioning, Disability and Health Model in Paediatric Cochlear Implant Recipients
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: ICF in Paediatric CI users
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cochlear Impant Children
MeSH Terms: interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cochlear Implant (CI) recipients (<18 years) with prelingual sensorineural hearing loss: Cochlear Implant (CI) recipients (<18 years) with prelingual sensorineural hearing loss
  Interventions: Device: Cochlear Implantation

INTERVENTIONS:
Device: Cochlear Implantation — Standard cochlear implantation

SUMMARY:
The aim of this study is to implement the International Classification of Functioning, disability and health (ICF) in paediatric Cochlear Implant (CI) recipients (<18 years) with prelingual sensorineural hearing loss in a multicenter prospective study to evaluate audiological rehabilitation after cochlear implantation. For this, ICF qualifiers which denote the magnitude of the level of health or severity of the problem will be quantified. Outcome measures include four questionnaires and three standard audiological examinations. Subjects will be assessed up to 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor.

ELIGIBILITY:
Inclusion Criteria:

General

* Children aged < 18 years with prelingual bilateral severe-to-profound HL
* Signed and dated informed consent, informed permission and/or minor's assent.
* Willingness to participate in evaluations, test sessions, and medical follow-up sessions as defined in the protocol.
* Physical and mental competence to participate in fitting of the device and follow-up sessions as defined in the protocol.

Audiological

* Completion of hearing assessment battery showing suitability of the CI candidates.
* Compliance with cochlear implant candidate selection criteria of the implanting centre.
* First cochlear implantation Medical
* Patent cochlea, as evidenced by High-resolution computed tomography (HRCT) and/or Magnetic Resonance Imaging (MRI).

Exclusion Criteria:

General

* Re-implantation of the cochlear implant
* No motivation to participate in the study and/or unreasonable expectations. Medical
* Presence of contra-indications for surgery in general and cochlear implantation in particular.
* Presence of central auditory lesions.
* Any disorder that may relate to an increased risk of skin flap problems Use of one of the following electrodes for implantation
* Compressed
* Split
* Any type of custom made electrodes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric Cochlear Implant (CI) recipients (<18 years) with prelingual sensorineural hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in LittlEARS® Auditory Questionnaire (LEAQ) | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  The LittlEARS® Auditory Questionnaire (LEAQ) was created to aid professionals and caregivers in the assessment of auditory capabilities among infants and toddlers experiencing hearing impairment. Grounded in the observations made by caregivers concerning the auditory responses exhibited by their children in everyday settings, this questionnaire comprises 35 questions tailored to specific age groups, necessitating responses of either 'yes' or 'no'. These questions are designed to capture significant milestones in auditory development during the initial two years of life or within the first two years following the onset of hearing intervention for children utilizing hearing devices. The questionnaire is suitable for children up to 24 months old, or with a hearing age of 24 months.
Change in Speech, Spatial and Qualities of Hearing Scale for Parents (SSQ-P) | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  The original SSQ was adapted for use in children, resulting in the development of the SSQ-P. Each of the 23 items in the questionnaire presents a scenario followed by a question regarding the child's hearing ability within that scenario. These items are categorized into three dimensions: speech perception, spatial hearing, and qualities of hearing. Parents are tasked with providing a rating between 0 and 10 for each item, where 0 signifies that the child could not perform in the scenario at all and 10 indicates perfect performance. Additionally, parents are asked to indicate how frequently the scenario would occur and to rate the importance of the listening skills required for that scenario.
Change in Speech Intelligibility Rating (SIR) | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  The Speech Intelligibility Rating (SIR) comprises spoken passages, wherein the degree of intelligibility is evaluated using an interval scale spanning from 0 to 10, ensuring uniformity in rating perception. The SIR assessment uses 20 standardized passages delivered by a single speaker, each identified as possessing comparable levels of intelligibility. The SIR is typically used in children with hearing loss from around the age of 2 years old .
Parent's Evaluation of Aural/Oral Performance of Children (PEACH) | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  The PEACH is a 13-item questionnaire designed for parental assessment of a 3- to 7-year-old child's aural and oral abilities in everyday life. The PEACH asks parents to consider their child's listening behaviors over the past week and then assigns a numerical value to the answers ranging from 0 (Never or 0 %) to 4 (Always or 75 to 100 %). The PEACH questions assess listening behaviors in both quiet and noisy surroundings.
Standard pure tone audiometry, Behavioral Observation Audiometry (BOA), Visual Reinforcement Audiometry (VRA) or Play Audiometry | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  Standard pure tone audiometry, Behavioral Observation Audiometry (BOA), Visual Reinforcement Audiometry (VRA) or Play Audiometry will be performed according to current clinical standards (ISO 8253-1, 2010), depending on the age of the participant. Pre- and postoperatively, best-aided audiometry will be measured at 250, 500, 1000, 2000, 4000 and 8000 Hz using warble tones in sound field in a sound treated booth. The loudspeaker will be placed in front of the participant at ear level at 1 meter distance. The best-aided pure tone average (PTA4, primary outcome measurement) will be calculated by averaging participants' hearing thresholds at 500, 1000, 2000 and 4000 Hz in best-aided condition.
Auditory Brainstem Response (ABR) Audiometry | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  ABR audiometry involves the generation of an evoked potential through a brief auditory stimulus (e.g., click, chirp, etc.) transmitted via an acoustic transducer (insert earphone or headphone). The resulting waveform response is detected by surface electrodes positioned at the vertex of the scalp and ear lobes. The signal's amplitude is averaged and plotted against time and waveform peaks are identified as I-VII. These waveforms typically occur within a 10-millisecond window following a click stimulus presented at high intensities (70-90 dB normal hearing level [nHL]). ABR audiometry is suitable for children of all ages.
Ling Sounds (detection/discrimination) | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  For Ling sound detection, the participants' detection of six sounds (oo, ah, ee, mm, sh, ss) will be observed in a variety of game formats. In the clinic, each sound is presented six times without lipreading, and the child simply responds. Score "S" will be given if the skill is emerging, score "A" will be given if the child has been observed to carry out the tasks consistently. For Ling discrimination, the phoneme "ee" will be repeated and all six Ling Sounds will be randomly inserted. Score "S" will be given if the child is consistently able to discriminate any one sound out of the six, score "A" will be given if the child is consistently able to discriminate all six sounds. The Ling test is suitable for children from approximately 6 months of age to adulthood.

SECONDARY OUTCOMES:
Subject Demographics | 1 month before implantation and 3 months, 6 months and 1 year post the activation of the speech processor
  Subject demographics will be retrieved from the participants' medical file or by asking the parents if the information is not available. The 11th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-11) classification will be used to code subjects' health conditions.

CONTACTS AND LOCATIONS:
Locations (6):
- Fiona Stanley Fremantle Hospital Group, Perth, Australia
- University Hospital Antwerp, Edegem, Belgium
- University Clinic of Würzburg, Würzburg, Germany
- World Hearing Centre, Warsaw, Poland
- King Abdullah Ear Specialist Center (KAESC), Riyadh, Saudi Arabia
- Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No